CLINICAL TRIAL: NCT05158894
Title: The Ubrelvy and Qulipta Pregnancy Exposure Registry EMPRESS: An Observational, Prospective Study to Assess the Safety of Ubrelvy (Ubrogepant) and Qulipta (Atogepant) During Pregnancy
Brief Title: Observational Study to Assess Adverse Events When Adult Female Participants Are Treated With Ubrelvy (Ubrogepant) or Qulipta (Atogepant) During Pregnancy
Acronym: EMPRESS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-392; MED-EPI-NEU-0649 (Other Grant/Funding Number: AbbVie)
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Migraine; Ubrelvy; Ubrogepant; Atogepant; Qulipta; MED-EPI-NEU-0649
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ubrelvy-Exposed Women With Migraine: Pregnant women with migraine who took at least 1 dose of Ubrelvy, the exposure of interest, at any time during pregnancy as part of routine care.
- Qulipta-Exposed Women With Migraine: Pregnant women with migraine who took at least 1 dose of Qulipta, the exposure of interest, at any time during pregnancy as part of routine care.
- Ubrelvy/Qulipta-Unexposed Women With Migraine: Pregnant women with migraine who have never taken Ubrelvy and/or Qulipta, OR discontinued Ubrelvy 2 days prior or Qulipta 5 days prior to conception.

SUMMARY:
Migraine is a common neurological disorder typically characterized by attacks of throbbing or pulsating headache on one side of the head of moderate to severe pain intensity. The purpose of this study is to evaluate fetal, maternal, and infant outcomes through 12 months of age among women exposed to Ubrelvy or Qulipta during pregnancy, as well as in 2 comparator groups.

Ubrelvy (ubrogepant) and Qulipta (atogepant) are approved drugs for the acute treatment of migraine in adults. Approximately 628 pregnant women with migraine exposed to Ubrelvy, 628 pregnant women with migraine exposed to Qulipta and 628 pregnant women with migraine in comparator group will be enrolled in this study in the United States.

Participants enrolled in the Ubrelvy-exposed group and Qulipta-exposed group will receive Ubrelvy and Qulipta respectively as prescribed by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Within the United States or Canada.
* Qualify as a prospective enrollment, defined as currently pregnant.
* A diagnosis of migraine by the patient's health care provider (HCP).
* Provide contact information for the participant and her and her infant(s)', if applicable, HCPs.
* Authorize their HCP(s) to release maternal and infant medical information to the registry, upon request.
* Provide sufficient information to confirm eligibility for 1 of following:

  * Ubrelvy-exposed women with migraine: documented information indicating that at least 1 dose of Ubrelvy was taken during pregnancy, including the estimated number of administrations per trimester.
  * Qulipta-exposed women with migraine: documented information to indicating that at least 1 dose of Qulipta was taken during pregnancy, including start and stop date(s) of administration.
  * Internal comparator: Ubrelvy/Qulipta-unexposed pregnant women with migraine: documented information indicating that they have, a) never taken Ubrelvy and/or Qulipta, or b) discontinued Ubrelvy 2 days prior or Qulipta 5 days prior to conception.

Exclusion Criteria:

* Documentation of exposure to any gepants (acute or preventive) other than Ubrelvy and Qulipta, or CGRP monoclonal antibodies, from 5 halflives of the respective treatment prior to conception or at any point during pregnancy before enrollment.
* Women who are no longer pregnant (retrospective cases women for whom the pregnancy has already ended, and the outcome of pregnancy is known at the time of enrollment).
* For further clarification of inclusion/exclusion please contact the investigator to the end of this section in case anything is unclear to a potential patient, etc

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of pregnant women, residing in the US and at least 18 years of age, and live born infants resulting from enrolled pregnancies. Participating women must meet eligibility criteria, including criteria for either the exposure or comparator group.
Sampling Method: Probability Sample
Enrollment: 1884 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Major Congenital Malformations (MCMs) | Up through the first 12 months of life
  An MCM is defined as any major structural or chromosomal defect in live born infants, stillbirths/fetal losses of any gestational age.

SECONDARY OUTCOMES:
Percentage of Pregnant Participants Experiencing Spontaneous Abortion | Up through the first 12 months of life
  Recognized spontaneous abortion (SAB): loss of an embryo/fetus due to natural causes prior to 20 weeks of gestation.
Percentage of Pregnant Participants Experiencing Stillbirth | Up through the first 12 months of life
  A fetal death occurring at 20 gestation weeks or greater, or if gestational age is unknown, a fetus weighing 350 g or more.
Percentage of Pregnant Participants With Elective Termination | Up through the first 12 months of life
  Elective termination is voluntary interruption of pregnancy, including pregnancy termination that occurs electively, to preserve maternal health, or due to abnormalities.
Percentage of Pregnant Participants Experiencing Preeclampsia | Up through the first 12 months of life
  Preeclampsia is the presence of hypertension on 2 occasions at least 4 hours apart after 20 weeks gestation (in a woman with a previously normal blood pressure) and proteinuria, or new-onset hypertension accompanied by thrombocytopenia, renal insufficiency, impaired liver function, pulmonary edema, or cerebral or visual symptoms.
Percentage of Pregnant Participants Experiencing Eclampsia | Up through the first 12 months of life
  Eclampsia is defined as new-onset seizures (tonic-clonic, focal, or multifocal) in the absence of other causative conditions such as epilepsy, cerebral arterial ischemia and infarction, intracranial hemorrhage, or drug use.
Percentage of Pregnant Participants Experiencing Gestational Hypertension | Up through the first 12 months of life
  Gestational hypertension is defined as high blood pressure (Elevated: systolic between 120-129 mm Hg and diastolic less than 80 mm Hg; Stage 1 hypertension: systolic between 130-139 mm Hg or diastolic between 80-89 mm Hg; Stage 2 hypertension: systolic at least 140 mm Hg or diastolic at least 90 mm Hg) associated with pregnancy.
Percentage of Pregnant Participants Experiencing Gestational Diabetes | Up through the first 12 months of life
  Gestational diabetes is generally characterized by the development of carbohydrate intolerance with first onset or first recognition during pregnancy; a record of an oral glucose tolerance test during pregnancy will also be accepted for data collection, where available.
Percentage of Infants Experiencing Preterm Birth | Up through the first 12 months of life
  Preterm birth is defined as an infant born at gestational age <37 weeks.
Percentage of Infants Experiencing Small for Gestational Age (SGA) Birth | Up through the first 12 months of life
  SGA at birth based on health care provider (HCP) report, typically defined as birthweight <=10th percentile for sex and gestational age.
Percentage of Infants Experiencing Minor Malformations | Up through the first 12 months of life
  Minor malformations not previously reported.
Percentage of Infants With Age-appropriate Infant Growth and Development | Up through the first 12 months of life
  Age-appropriate progress on developmental milestones based on the overall assessment by the infant's HCP (e.g., appropriate or delayed) up to 1 year of age.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- Iqvia /Id# 266904, Durham, North Carolina, United States
- Ottawa Hospital Research Institute /ID# 280174, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.empresspregnancyregistry.com